CLINICAL TRIAL: NCT00984061
Title: A Pharmacokinetic Study to Evaluate the Effect of Clarithromycin on the Pharmacokinetic Profile of Colchicine in Healthy Adults
Brief Title: Drug-Drug Interaction Study of Colchicine and Clarithromycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-07-1006
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
Keywords: healthy; pharmacokinetics; drug-drug interaction
MeSH Terms: interventions — Colchicine; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- colchicine alone (Experimental): colchicine baseline pharmacokinetics
  Interventions: Drug: colchicine
- colchicine with clarithromycin (Experimental): colchicine pharmacokinetics in presence of clarithromycin
  Interventions: Drug: clarithromycin; Drug: colchicine

INTERVENTIONS:
Drug: colchicine — 0.6mg tablet administered at 9am on Day 1
  Arms: colchicine alone
Drug: clarithromycin — 250 mg clarithromycin tablet taken on an outpatient basis twice daily at 8am and 8pm for 14 doses (starting with 8pm dose on Day 22 and concluding with 8am dose on Day 29)
  Arms: colchicine with clarithromycin
Drug: colchicine — 0.6 mg tablet administered at 9am on Day 29
  Arms: colchicine with clarithromycin

SUMMARY:
Clarithromycin is a potent inhibitor of the activity of cytochrome P450 (CYP) 3A4 and P-glycoprotein (P-gp). CYP 3A4 plays a role in the metabolism of colchicine and P-gp is responsible for the efflux of colchicine across membranes. This study will evaluate the effect of clarithromycin-related inhibition of CYP 3A4 and P-gp on the pharmacokinetics of colchicine. It will also evaluate the safety and tolerability of concurrent administration of clarithromycin and a single dose of colchicine.

DETAILED DESCRIPTION:
Clarithromycin is a potent inhibitor of the activity of cytochrome P450 (CYP) 3A4 and P-glycoprotein (P-gp). CYP 3A4 plays a role in the metabolism of colchicine and P-gp is responsible for the efflux of colchicine across membranes. This open-label, one sequence, two-period, drug-drug interaction study will evaluate the effect of clarithromycin-related inhibition of CYP 3A4 and P-gp on colchicine pharmacokinetics in 24 healthy, non-smoking, non-obese (within +/- 15% of ideal body weight), male and female adult volunteers. The safety and tolerability of concurrent administration of clarithromycin and a single dose of colchicine will also be evaluated. During the first period, subjects will be confined to the study unit beginning the afternoon of the day prior to scheduled dosing (Day -1). On the morning of Day 1, after an overnight fast of at least 10 hours, subjects will be administered a single dose of colchicine 0.6 mg tablet with 240 ml of room temperature water. Blood will be drawn at times sufficient to characterize the baseline pharmacokinetics for this group. Following a 20 day washout period on Day 22, all subjects will return to the clinic to receive a supply of clarithromycin 250 mg tablets, which they will take on an outpatient basis twice daily (at 8 a.m. and 8 p.m.) without regard to meals for a total of 14 doses. Clinic staff will make telephone contact daily with subjects during this course to confirm compliance with the clarithromycin dosing regimen, and to monitor for adverse events and use of concomitant medication. On day 28 in the afternoon, subjects will again be confined to the study unit. On the morning of day 29, after an overnight fast of at least 10 hours all subjects will be administered a single dose of colchicine 0.6 mg and the final dose of clarithromycin with 240 ml water. Blood samples will be drawn at times sufficient to determine pharmacokinetic profiles of colchicine in the presence of clarithromycin at steady state. The pharmacokinetic profiles will be compared to determine the extent of drug-drug interaction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, adult volunteers, male and female, 18 to 45 years of age, weighing at least 55 kg and within 15% of ideal body weight, with hemoglobin >/=12 g/dL.
* Female volunteers must be sexually abstinent for 14 days prior to the first dose and throughout the study or using acceptable birth control methods (prior to and during the study), including being postmenopausal or surgically sterile (or sexual activity restricted to a partner that is surgically sterile), hormonal contraception, an IUD, or barrier methods with spermicide. Additionally, they will be advised to remain sexually inactive or to keep the same birth control method for at least 14 days following the last dose of colchicine.

Exclusion Criteria:

* Subjects who are pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg) or hepatitis C virus (HCV)
* Have history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease; have used any drugs or substances known to inhibit or induce CYP enzymes and/or P-gp within 30 days prior to the first dose and throughout the study
* Recent (2-year) history of evidence of alcoholism or drug abuse
* Subjects who donated 50-499 ml of blood within 30 days and more than 499 ml within 56 days prior to the first dose; subjects who have donated in excess of 500 ml of blood in 14 days, 1500 ml or blood in 180 days, or 2500 ml of blood in 1 year (through completion of the study)
* Have participated in another clinical trial within 30 days prior to dosing
* Known and documented drug allergies to colchicine or macrolide antibiotics.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Study Chair — Mutual Pharmaceutical Company, Inc.
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking, adult male and female volunteers, consisting of members of the community at large, were enrolled.
Pre-assignment Details: 56 subjects screened, 32 were screen failures
Groups:
- Colchicine Alone / With Clarithromycin: [All subjects received each of the study treatments.] Each subject received one colchicine 0.6 mg tablet on Day 1 at 9:00 a.m. after an overnight fast of at least 10 hours, followed by a 21 day washout period. On Day 22, subjects began taking one 250 mg clarithromycin tablet every 12 hours at 8:00 a.m. and 8:00 p.m. for 7 days without regard to meals. Then, on Day 29, each subject received one colchicine 0.6 mg tablet along with final dose of 250 mg clarithromycin at 9:00 a.m. after an overnight fast of at least 10 hours.
Period: Colchicine Alone
Arm/Group | Colchicine Alone / With Clarithromycin
Started | 24
Completed | 24
Not Completed | 0
Period: 21 Day Washout Period
Arm/Group | Colchicine Alone / With Clarithromycin
Started | 24
Completed | 24
Not Completed | 0
Period: Clarithromycin Alone
Arm/Group | Colchicine Alone / With Clarithromycin
Started | 24
Completed | 23 (One subject was dropped due to noncompliance with outpatient clarithromycin regimen.)
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Colchicine With Clarithromycin
Arm/Group | Colchicine Alone / With Clarithromycin
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine Alone / With Clarithromycin
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — age range: >=18 and <=45 years old
  Participants
    <=18 years | 0
    Between 18 and 65 years | 24
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.3 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 24
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples collected immediately prior to dosing on Days 1 and 29, then at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours after dose administration
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Colchicine Alone: Each subject received one colchicine 0.6 mg tablet on Day 1 at 9:00 a.m. after an overnight fast of at least 10 hours, followed by a 21 day washout period.
- Colchicine With Clarithromycin: On Day 22, subjects began taking one 250 mg clarithromycin tablet every 12 hours at 8:00 a.m. and 8:00 p.m. for 7 days without regard to meals. Then, on Day 29, each subject received one colchicine 0.6 mg tablet along with final dose of 250 mg clarithromycin at 9:00 a.m. after an overnight fast of at least 10 hours.
Arm/Group | Colchicine Alone | Colchicine With Clarithromycin
Number analyzed (Participants) | 23 | 23
ng/mL | 2.84 (0.88) | 8.44 (1.49)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the colchicine plasma concentration versus time curve beginning from the first dose (time 0) to the last measurable colchicine concentration (time t), as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Clarithromycin
Number analyzed (Participants) | 23 | 23
ng-hr/mL | 12.37 (4.66) | 41.95 (9.78)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the colchicine plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Clarithromycin
Number analyzed (Participants) | 23 | 23
ng-hr/mL | 15.53 (7.70) | 52.62 (12.02)

ADVERSE EVENTS:
Groups:
- Colchicine Alone: On the morning of Day 1 after a fast of at least 10 hours, all subjects received a single dose of colchicine 0.6 mg.
- Clarithromycin Alone: On the evening of Day 22, subjects began taking (on an outpatient basis) one tablet of clarithromycin 250 mg every 12 hours for 7 days without regard to meals.
- Colchicine With Clarithromycin: On the morning of Day 29 after an overnight fast of at least 10 hours, all subjects received a single dose of colchicine 0.6 mg along with the last dose of clarithromycin.
Arm/Group | Colchicine Alone | Clarithromycin Alone | Colchicine With Clarithromycin
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 7 | 5 | 4
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Alone | Clarithromycin Alone | Colchicine With Clarithromycin
hypoacusis (Ear and labyrinth disorders) | 1/24 (1) | 0/23 (0) | 0/23 (0)
abdominal pain upper (Gastrointestinal disorders) | 0/24 (0) | 1/23 (1) | 0/23 (0)
diarrhea (Gastrointestinal disorders) | 0/24 (0) | 0/23 (0) | 2/23 (2)
nausea (Gastrointestinal disorders) | 2/24 (2) | 0/23 (0) | 2/23 (2)
stomach discomfort (Gastrointestinal disorders) | 0/24 (0) | 1/23 (1) | 0/23 (0)
chest pain (General disorders) | 0/24 (0) | 0/23 (0) | 1/23 (1)
vessel puncture site hematoma (General disorders) | 1/24 (1) | 0/23 (0) | 0/23 (0)
skin laceration (Injury, poisoning and procedural complications) | 1/24 (1) | 0/23 (0) | 0/23 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2/24 (2) | 1/23 (2) | 0/23 (0)
dizziness (Nervous system disorders) | 1/24 (1) | 0/23 (0) | 0/23 (0)
headache (Nervous system disorders) | 3/24 (4) | 2/23 (2) | 2/23 (2)
syncope (Nervous system disorders) | 2/24 (2) | 0/23 (0) | 0/23 (0)
vision blurred (Nervous system disorders) | 1/24 (2) | 0/23 (0) | 1/23 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 1/23 (1) | 0/23 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/24 (1) | 0/23 (0) | 0/23 (0)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 1/23 (1) | 0/23 (0)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1/24 (1) | 0/23 (0) | 0/23 (0)
pallor (Vascular disorders) | 2/24 (2) | 0/23 (0) | 0/23 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days